CLINICAL TRIAL: NCT05875493
Title: A Phase I, Single-center, Randomized, Open-label, 2-cycle,2-period Crossover Study to Evaluate the Food Effect on the Pharmacokinetics of JAB-21822 in Healthy Subjects
Brief Title: A Food Effect Study of JAB-21822 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JAB-21822-1009
Record Dates: First submitted 2023-04-23; First posted 2023-05-25 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-01

CONDITIONS: Food Effect in Healthy Participants

STUDY DESIGN:
Intervention Model Description: This is an open-label,randomized, 2-cycle,2-period crossover,food effect study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A-JAB-21822 (Experimental): Dosing in the fasted state followed by fed dosing
  Interventions: Drug: JAB-21822
- B-JAB-21822 (Experimental): Dosing in the fed state followed by fasted dosing
  Interventions: Drug: JAB-21822

INTERVENTIONS:
Drug: JAB-21822 — 2 discrete single doses
  Arms: A-JAB-21822
Drug: JAB-21822 — 2 discrete single doses
  Arms: B-JAB-21822

SUMMARY:
The primary objective of this study is to determine the effect of food in healthy participants on the bioavailability of JAB-21822 following single dose administration with and without a meal

DETAILED DESCRIPTION:
This is an open-label,randomized, 2-cycle,2-period crossover,food effect study. On Day 1 of each period, subjects will receive a single oral dose of JAB-21822 administered either under fasting conditions or following a standardized high-fat/high-calorie meal. PK sampling for JAB-21822 will be collected predose and postdose. There will be a washout period between doses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female , between 18 and 45 years of age
* Bodyweight (male) ≥50kg, Bodyweight (Female) ≥45kg；BMI within the range of 19 to 25 kg/m2, inclusive
* No clinically significant abnormalities identified in the judgement of investigator at screening
* Written informed consent prior to any study specific procedures

Exclusion Criteria:

* History of clinically significant disease or disorder
* History of interstitial pneumonia, pulmonary fibrosis, and other interstitial lung diseases
* History of dysphagia or any gastrointestinal disease that would potentially alter absorption of drug
* COVID-19 positive at screening or baseline
* Allergic to JAB-21822 and any of the tablet's ingredients, history of hypersensitivity or allergy to drug or food
* Received surgical procedure within 3 months at screening
* Blood donation within the 3 months or planing to donate during the study
* Participated in another clinical trial of biological agents within 6 months at screening, or any other clinical trial within 3 months at screening
* History of drug abuse or positive urine drug test
* Received the vaccine within 3 months at screening or planning to receive during the study
* Overtake of achole,tea and coffee prior to first dosing and unable to control during the study
* Special dietary requirements or unable to control during the study
* HIV, HBV, HCV, and syphilis positive
* Pregnant or breast-feeding women or positive of blood pregnancy test
* Subjects who are considered to be unacceptable in this study under the opinion of the investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration (AUC) 0 to∞ | 31days
  Area under the plasma concentration time curve of JAB-21822
Area under plasma concentration (AUC) 0 to t | 31days
  Area under the plasma concentration time curve of JAB-21822
Plasma concentration ( Cmax) | 31days
  Highest observed plasma concentration of JAB-21822

SECONDARY OUTCOMES:
Time to achieve Cmax (Tmax) | 31days
  Time of highest observed plasma concentration of JAB-21822
Elimination rate constant (λz) | 31days
  Elimination rate constant based on the terminal phase of unchanged form of JAB-21822
Concentration half-life (T1/2) | 31days
  Elimination half-life of unchanged form of JAB-21822
Absorption lag-time (Tlag) | 31days
  Elimination lag-time of JAB-21822
Apparent volume of distribution (Vz/F) | 31days
  Apparent volume of distribution based on the terminal phase of unchanged form of JAB-21822
Apparent clearance (CL/F) | 31days
  Apparent total body clearance of unchanged form of JAB-21822
Number of participants with adverse events (AEs) and serious adverse events(SAEs) | 31days
  Incidence,duration and severity of adverse events and serious adverse events according to NCI-CTCAE v5.0
Number of subjects with abnormal lab parameters | 31days
  Abnormal values of lab parameters
Number of subjects with abnormal electrocardiogram (12-lead ECG) | 31days
  Prolongation of the QTc interval
Number of subjects with abnormal systolic and diastolic blood pressure | 31days
  Abnormal values in systolic and diastolic blood pressure
Number of subjects with abnormal pulse rate | 31days
  Abnormal values in pulse rate
Number of subjects with abnormal respiratory rate | 31days
  Abnormal values in respiratory rate
Number of subjects with abnormal body temperature | 31days
  Abnormal values of body temperature

CONTACTS AND LOCATIONS:
Overall Officials: He Qing B.Pharm, Principal Investigator — Beijing Gaobo Boren Hospital
Locations (1):
- Beijing GoBroad Boren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No